CLINICAL TRIAL: NCT06549413
Title: 18F-FSPG PET/CT as a Non-Invasive Imaging Biomarker for Treatment Response to Chemoradiation in Esophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0989; NCI-2023-04988 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2022-0989 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients receive 18F-FSPG IV and undergo a PET/CT scan. During week 3 of standard of care radiation therapy, patients receive 18F-FSPG and undergo a second PET/CT scan on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to learn how 18F-FSPG PET/CT scan results may be related to the response to chemotherapy and radiation in patients with esophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the ability of 18F-FSPG PET imaging to detect tumors in patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* * ≥ 18 years of age

  * Patients with locally advanced esophageal cancer
  * Patients with untreated documented carcinoma of the esophagus that is > 2 cm who are going to receive systemic therapy concurrently with radiation as primary therapy
  * Ability to provide written informed consent in accordance with institutional policies
  * Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 1 week of the proposed investigational PET/CT scan(s) prior to injection of the investigational radiopharmaceutical

Exclusion Criteria:

* * Body weight ≥ 400 pounds or body habitus or disability that will not permit the imaging protocol to be performed

  * Pregnant or lactating females
  * Have an allergy to intravenous contrast
  * eGFR < 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced esophageal cancer being seen at the Thoracic Radiation Oncology Section at the University of Texas MD Anderson Cancer Center (MDACC).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org